CLINICAL TRIAL: NCT04124952
Title: Evaluation of Quality of Vision and Spectacle Independence With Bilateral Implantation of the AcrySof® Panoptix® Intraocular Lens
Brief Title: Evaluation of Quality of Vision and Spectacle Independence With the AcrySof® Panoptix® Intraocular Lens
Status: Completed | Type: Observational
Sponsor: SightTrust Eye Institute (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Other Study IDs: AS-19-001
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2021-08

CONDITIONS: Cataract
Keywords: Panoptix, trifocal IOL, multifocal IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Panoptix: Patients bilaterally implanted with the Panoptix intraocular lens.
  Interventions: Device: Panoptix

INTERVENTIONS:
Device: Panoptix — Alcon Acrysof(R) Panoptix(R) intraocular lens (IOL)

SUMMARY:
This is a study to assess the spectacle independence and quality of vision of patients receiving the AcrySof® Panoptix® Intraocular lens (IOL) after uneventful cataract surgery.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of spectacle independence after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 day, 1 month and 3 months post-operatively. Clinical evaluations will include administration of a spectacle independence questionnaire, as well as measurement of bilateral visual acuity and manifest refraction.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Presenting for uncomplicated bilateral cataract surgery and have an interest in spectacle independence using a multifocal IOL or multifocal toric IOL option
* Gender: Males and Females.
* Age: 40 or older.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract)
* Have regular corneal astigmatism with a magnitude that can be treated with a non-toric IOL or a toric IOL in the approved ranged for the Panoptix lens.
* Have 20/32 (0.2 logMAR) or better potential acuity in both eyes

Exclusion Criteria If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Irregular astigmatism (e.g. keratoconus)
* Corneal pathology (e.g. scar, dystrophy, pterygium, severe dry eye)
* Monocular status (e.g. amblyopia)
* Previous radial keratotomy, corneal refractive surgery or other corneal surgery (e.g. corneal transplant, lamellar keratoplasty)
* Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy)
* Diabetic retinopathy
* Macular pathology (e.g. age-related macular degeneration, epiretinal membrane)
* History of retinal detachment
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity.
* Participation in any investigational drug or device trial within the previous 30 days prior to the start date of this trial (or currently participating).

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects ≥40 years of age presenting for cataract surgery who are interested in reducing their dependence on spectacles at all distances, and who are appropriate candidates for multifocal lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Shatz, MD, Principal Investigator — SightTrust Eye Institute
Locations (1):
- SightTrust Eye Institute, Sunrise, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
No current plans exist. If data are shared, they will be de-identified beforehand.

REFERENCES:
- [Background] Morlock R, Wirth RJ, Tally SR, Garufis C, Heichel CWD. Patient-Reported Spectacle Independence Questionnaire (PRSIQ): Development and Validation. Am J Ophthalmol. 2017 Jun;178:101-114. doi: 10.1016/j.ajo.2017.03.018. Epub 2017 Mar 22. PMID 28341605
- [Background] McAlinden C, Pesudovs K, Moore JE. The development of an instrument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5537-45. doi: 10.1167/iovs.10-5341. Epub 2010 May 26. PMID 20505205

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Panoptix
Started | 30
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were for subjects completing the study
Arm/Group | Panoptix
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Emmetropic Subjects Who Are Spectacle Independent
Description: Number of patients who have a 3-month postoperative manifest spherical equivalent refraction within 0.5 diopters (D) of plano, and ≤ 0.5 D of refractive cylinder (emmetropic subgroup) who never or rarely wear spectacles for distance, intermediate or near vision 3 months postop (based on the Patient-Reported Spectacle Independence Questionnaire (PRSIQ) - "a little of the time" or "none of the time").
Time Frame: 3 months
Population: This is the number of emmetropic subjects (subgroup)
Measure: Count of Participants; unit: Participants
Arm/Group | Panoptix
Number analyzed (Participants) | 21
Participants | 21

2. Secondary Outcome: Binocular Uncorrected Distance Visual Acuity
Description: Binocular logMAR uncorrected distance visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Panoptix
Number analyzed (Participants) | 29
logMAR | 0.07 (0.09)

3. Secondary Outcome: Binocular Uncorrected Intermediate Visual Acuity
Description: Binocular logMAR uncorrected intermediate visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Panoptix
Number analyzed (Participants) | 29
logMAR | 0.09 (0.13)

4. Secondary Outcome: Binocular Uncorrected Near Visual Acuity
Description: Binocular logMAR uncorrected near visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR Acuity
Arm/Group | Panoptix
Number analyzed (Participants) | 29
logMAR Acuity | 0.07 (0.11)

5. Secondary Outcome: Binocular Corrected Distance Visual Acuity
Description: Binocular logMAR corrected distance visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR Acuity
Arm/Group | Panoptix
Number analyzed (Participants) | 29
logMAR Acuity | 0.03 (0.07)

6. Secondary Outcome: Binocular Distance-corrected Intermediate Visual Acuity
Description: Binocular distance-corrected intermediate visual acuity in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR Acuity
Arm/Group | Panoptix
Number analyzed (Participants) | 29
logMAR Acuity | 0.06 (0.10)

7. Secondary Outcome: Binocular Distance-corrected Near Visual Acuity
Description: Binocular logMAR distance-corrected near visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR Acuity
Arm/Group | Panoptix
Number analyzed (Participants) | 29
logMAR Acuity | 0.05 (0.11)

8. Secondary Outcome: Spherical Equivalent Refraction
Description: Spherical equivalent refraction in diopters
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Panoptix
Number analyzed (Participants) | 29
diopters | 0.06 (0.53)

9. Secondary Outcome: Residual Refractive Cylinder
Description: Residual refractive cylinder in diopters
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Panoptix
Number analyzed (Participants) | 29
diopters | 0.49 (0.36)

10. Secondary Outcome: Quality of Vision Questionnaire
Description: Quality of Vision questionnaire results. This is a Rasch-scaled test with scores from 0-100, with lower being better.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Score on a scale (0-100, 0 is best)
Arm/Group | Panoptix
Number analyzed (Participants) | 29
Score on a scale (0-100, 0 is best)
  Frequency | 36.9 (16.6)
  Severity | 30.6 (15.1)
  Degree of bother | 28.7 (20.7)

11. Secondary Outcome: Overall Spectacle Independence
Description: percent of all patients who never or rarely wear spectacles for distance, intermediate or near vision 3 months postop (based on the PRSIQ - "a little of the time" or "none of the time")
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Panoptix
Number analyzed (Participants) | 29
Participants | 29

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Panoptix
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panoptix (N=30)
Bicycle accident (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT04124952/Prot_SAP_000.pdf